CLINICAL TRIAL: NCT06025708
Title: Impact of Sample Type on the Performance of the Quantra QStat System
Brief Title: Quantra QStat Sample Type Comparison
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-046
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Coagulation Defect; Bleeding
Keywords: Quantra; Liver transplantation; Coagulation
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Diagnostic Test: Quantra QStat Cartridge — Whole blood coagulation testing system

SUMMARY:
This is a single center prospective observational study to compare QStat parameter measurements in arterial and venous blood samples collected in parallel from patients undergoing liver transplantation.

DETAILED DESCRIPTION:
In this single center prospective observational study, 25 cardiac surgery subjects will enrolled, each with parallel artrial and venous samples collected at 3 time points to yield 75 matched samples for analysis on the Quantra System with the QStat Cartridge.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >=18 years
* Subject is scheduled for liver transplant surgery
* Subject or subject's legally authorized representative (LAR) is willing to provide informed consent

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject is pregnant
* Subject is incarcerated at the time of the study
* Subject is affected by a condition that, in the opinion of the treatment team, may pose additional risks
* Subject, or subject's LAR, is unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing liver transplant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of QStat Clot time (CT) in arterial and venous samples | During liver transplantation surgery
  Coagulation function assessed in two sample types
Comparison of QStat Clot stiffness (CS) in arterial and venous samples | During liver transplantation surgery
  Coagulation function assessed in two sample types
Comparison of QStat Platelet Contribution to Clot stiffness (PCS) in arterial and venous samples | During liver transplantation surgery
  Coagulation function assessed in two sample types
Comparison of QStat Fibrinogen Contribution to Clot stiffness (FCS) in arterial and venous samples | During liver transplantation surgery
  Coagulation function assessed in two sample types
Comparison of QStat Clot Stabilty to Lysis (CSL) in arterial and venous samples | During liver transplantation surgery
  Coagulation function assessed in two sample types

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No